CLINICAL TRIAL: NCT00690274
Title: A Randomized, Double Blind, Placebo Controlled, Study to Demonstrate the Cognitive Enhancing Effects of BF2.649 in People With Schizophrenia and Schizoaffective Disorder
Brief Title: Study to Demonstrate Cognitive Enhancing Effects of BF2.649
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Bioprojet (Other); Stanley Medical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BF2.649
Record Dates: First submitted 2008-06-02; First posted 2008-06-04 (Estimated); Results first posted 2019-04-23 (Actual); Last update posted 2019-04-23 (Actual); Status verified 2019-03

CONDITIONS: Schizophrenia
Keywords: schizophrenia; cognitive deficients; cognitive enhancing; antipsychotics
MeSH Terms: conditions — Schizophrenia | interventions — pitolisant; Starch

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Volunteers are given Placebo, up to 20mg per day
  Interventions: Drug: Placebo
- BF2.649 (Active Comparator): Volunteers are given BF2.649, up to 20mg per day
  Interventions: Drug: BF2.649

INTERVENTIONS:
Drug: BF2.649 — up to 20mg per day
  Other Names: Study medication
  Arms: BF2.649
Drug: Placebo — up to 20mg per day
  Other Names: cornstarch capsule
  Arms: Placebo

SUMMARY:
To evaluate the cognitive enhancing effect of BF2.649 and to evaluate the effect of BF2.649 on symptom severity in persons with schizophrenia or schizoaffective disorder.

DETAILED DESCRIPTION:
We will recruit persons with schizophrenia or schizoaffective disorder who are not currently experiencing an acute exacerbation of psychotic symptoms, but still display cognitive symptoms and have consequent psychosocial dysfunction. The subjects recruited will be taking haloperidol, aripiprazole, risperidone or paliperidone. Each study subject will spend 4 weeks on a fixed dose of his or her APD with stable symptoms, during which time the baseline workup will be completed. At baseline (Week 0), each study subject will have a full symptom evaluation, side effects, and neuropsychological battery along with the full clinical laboratory and baseline safety study workup. Next, subjects, while remaining on their APD, will be randomized to BF2.649 or placebo. The dose of BF2.649 will be up to 20 mg/day. Assessment of safety parameters (vital signs, EKGs, clinical labs) and side effects (adverse events, BAS, SAS) will occur once weekly for the first 4 weeks (through study week 4) and then every other week for the next 4 weeks (to study week 8) including End of Study (week 12). An EEG will be taken at Week 1 and then at Week 8. Symptomatic outcome measures (PANSS and CGI) will be measured every two weeks during the double blind phase and at end of study. The neuropsychological battery will be done first at baseline and repeated at the end of the 8-week double blind phase. After 8 weeks of medication, the double-blinded drug will be stopped and the patient followed for a period 4 weeks with clinical and side effect measures recorded weekly with the exception of clinical laboratories, which will be recorded every other week. Each study participant will be seen weekly throughout the protocol for clinical assessment.

Finally, persons with schizophrenia display severe deficits in neuropsychological, cognitive, and social functioning. Our primary outcome measure will be to determine if BF2.649 can produce a cognitive enhancing effect and repair some of the neuropsychological deficiencies seen in this population. Therefore, blood samples will be collected from study volunteers for DNA analysis, serology testing, and white cell immortalization during and only at the baseline phase of the study (Week 0). If a therapeutic effect is seen, it will be important to be able to identify the genetic characteristics of the responders to BF2.649.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV diagnosis of schizophrenia and schizoaffective disorder and not experiencing an acute exacerbation of severe psychosis
* Stable antipsychotic drug treatment for at least 4 weeks of Abilify or Haldol or willing to switch to either of these two APDs.
* Able to execute written informed consent.
* Males and females, between the ages of 18-55 years old, in good health (based on medical history, physical examination, electrocardiograms, and clinical laboratory tests)
* All races and ethnicities fluent and literate in English.

Exclusion Criteria:

* Diagnosis of DSM-IV alcohol or substance abuse within the last month or DSM-IV alcohol or substance dependence within the last 3 months.
* Patients on a stable regimen of antipsychotic medication (other than Haldol or Abilify) for a minimum of 3 months who are not experiencing psychotic symptoms.
* Clinically significant abnormal pre-admission vital signs, EKGs, or clinical laboratory evaluations, in which the principle investigator deems the subject-volunteer ineligible for the study.
* Any patient scheduled to undergo any surgical procedure during the duration of the study
* Patients suffering an acute psychotic episode within the previous 30 days as determined by the attending physician or Principal Investigator.
* Patients on any antihistaminergic antipsychotic medications who are not willing to switch to either Haldol or Abilify.
* Any patient who has received any known hepatic or renal clearance altering agents (e.g., erythromycin, cimetidine, barbiturates, phenothiazines, etc.) for a period of 3 months before the first dose of study medication
* Patients taking any concurrent medications for a major medical illness.
* Any patients who test positive for HIV.
* Any patient testing positive for Hepatitis B or C whose liver panel (taken during clinical laboratories) reports clinically significant abnormalities of liver enzyme ranges suggesting a cirrhotic stage.
* Any patient who has donated plasma or blood within 30 days before the first dose of study medication
* Concurrent treatment with electroconvulsive therapy.
* Pregnant women, women in the child bearing age without an efficacious contraceptive device, or women who are breast feeding.
* Mental capacity is limited to the extent that the patient cannot provide legal consent or understand information regarding the side effects or tolerance of the study drug
* Any patient judged by the principal investigator to be inappropriate for the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2008-06; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carol A Tamminga, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (2):
- United States (2):
  - UT Southwestern Medical Center, Dallas, Texas
  - The University of Texas Southwestern Medical Center, Dallas, Texas

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | BF2.649
Started | 29 | 23
Completed | 23 | 15
Not Completed | 6 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | BF2.649 | Total
Number analyzed (Participants) | 23 | 15 | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 23 | 15 | 38
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 11 | 29
  Male | 5 | 4 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 23 | 14 | 37
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 5 | 10
  White | 18 | 10 | 28
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 23 | 15 | 38

OUTCOME MEASURES:

1. Primary Outcome: Changes in Delayed Recall From Baseline to 12 Weeks
Description: The Brief Visuospatial Memory Test-Revised (Delayed Recall) is a neuropsychological test to assess one's ability to recall a previously exposed stimuli. The t-score range (as being reported) is from 35-81, with higher scores being better and indicating being able to recall more items after a 45-minute delay. (The t-score is a score calculated from the individual score and based on each individual's age group.) The t-scores are then grouped together and reported as a mean with the standard deviation.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: t-score
Arm/Group | Placebo | BF2.649
Number analyzed (Participants) | 23 | 15
t-score | 40.2 (2.9) | 43.4 (3.5)

2. Secondary Outcome: To Evaluate the Effect of BF2.649 on Symptom Severity Between Baseline and Week 12
Description: Montgomery-Asberg Depression Rating Scale (MADRS), a depression rating scale. The score can total from 0-60, with the higher score indicating more severe depressive symptoms. The scores indicate a change between baseline and 12 weeks.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | BF2.649
Number analyzed (Participants) | 23 | 15
scores on a scale | 0.5 (1.5) | -4.9 (1.9)

ADVERSE EVENTS:
Arm/Group | Placebo | BF2.649
Serious Adverse Events (participants affected / at risk) | 0/23 | 1/15
Other Adverse Events (participants affected / at risk) | 0/23 | 0/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=23) | BF2.649 (N=15)
suicidality (Psychiatric disorders) | 0 (0) | 1 (1) — Participant was expressing suicidal ideation and was psychiatrically hospitalized for evaluation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No